CLINICAL TRIAL: NCT01339169
Title: A Single Centre, Pilot Trial of YF476 in Patients With Chronic Atrophic Gastritis, Hypergastrinaemia and Type I Gastric Carcinoids
Brief Title: YF476 and Type I Gastric Carcinoids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trio Medicines Ltd. (Industry)
Collaborators: Royal Liverpool University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-008; 2007-002916-24 (EudraCT Number)
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Chronic Atrophic Gastritis; Hypergastrinaemia; Type I Gastric Carcinoids
Keywords: YF476; Hypergastrinaemia; netazepide; gastric carcinoids
MeSH Terms: conditions — Gastritis, Atrophic | interventions — YF 476

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YF476 treatment (Experimental)
  Interventions: Drug: YF476

INTERVENTIONS:
Drug: YF476 — 50 mg once daily for 12 weeks, with the option to increase to 75 mg or 100 mg once daily after 6 weeks, or decrease to 25 mg once daily, depending on response. After that, patients that have benefited from treatment may take 50 mg YF476 once daily for an additional up to 52 weeks.
  Other Names: netazepide

SUMMARY:
The aim of the study is to find out if the experimental medicine, YF476, can make gastric carcinoids, a rare type of stomach tumour, shrink and disappear. Gastric carcinoids occur mainly in patients with chronic atrophic gastritis (CAG), a condition in which the acid-producing cells in the lining of the stomach can't make acid. Acid production is controlled by gastrin, a hormone (chemical messenger) that's released into the bloodstream. If the stomach can't make acid, blood levels of gastrin rise. High blood levels of gastrin in patients with CAG can cause other cells (ECL cells) in the lining of the stomach to grow and, over the years, to give rise to gastric carcinoids. Gastric carcinoids are usually benign, but they can become malignant. Therefore, patients with CAG and gastric carcinoids have the inside of their stomach checked regularly, by gastroscopy, to see if the gastric carcinoids need removing surgically. A gastroscope is a thin (1 cm), flexible tube at end of which is a mini video camera, which enables the user to inspect the lining of the stomach and a 'snare' to take samples of tissue (biopsies). YF476 (netazepide) is a gastrin receptor antagonist (blocks the effects of gastrin), so it's a potential new medical treatment for gastric carcinoids in patients with CAG. Up to 10 of these patients will take YF476 daily for up to 12 weeks. If they benefit from that treatment, they may take YF476 daily for up to another 52 weeks. They'll make several outpatient visits for tests, including checks on the safety of YF476. At some of the visits, they'll have a gastroscopy. At each gastroscopy, the gastric carcinoids will be measured and biopsies taken for laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients known to have gastric carcinoids associated with chronic atrophic gastritis and hypergastrinaemia, and who attend the outpatient clinic of the investigator;
* Men, postmenopausal women, premenopausal women who have been sterilised by tubal ligation, hysterectomy or bilateral oophrectomy, or premenopausal women using reliable contraception: condom and spermicide or intrauterine device;
* Adults ≥ 18 years;
* Good general health; and
* Able to give fully-informed, written consent.

Exclusion Criteria:

* Women who are pregnant, lactating or using a steroid contraceptive;
* History of gastric surgery, apart from surgery for gastric carcinoids;
* Evidence of Zollinger-Ellison syndrome;
* Prolonged QTc interval (>450 msec);
* Certain medicines and herbal remedies taken during the 7 days before visit 1;
* Previous treatment with somatostatin; or
* Participation in other clinical trials of unlicensed medicines within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-01-04 (Actual); Primary Completion 2013-12-10 (Actual); Study Completion 2013-12-10 (Actual)

PRIMARY OUTCOMES:
Visual assessment of the number of gastric carcinoids. | 2 years
Visual assessment of the size of gastric carcinoids. | 2 Years
Visual assessment of the distribution of gastric carcinoids. | 2 years

SECONDARY OUTCOMES:
Safety and tolerability of YF476, as judged by medical examinations, vital signs, ECG, safety tests of blood and urine, and adverse events. | 2 years
Histologic grading of biopsies. | 2 years
Plasma concentrations of YF476. | 2 years
Plasma or serum concentrations of biomarkers such as gastrin or chromogranin A (CgA). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Boyce, BSc FRCP FFPM, Study Director — Trio Medicines Ltd.; Mark Pritchard, PhD FRCP, Principal Investigator — Royal Liverpool University Hospital
Locations (1):
- Royal Liverpool University Hospital, Liverpool, United Kingdom

REFERENCES:
- [Derived] Moore AR, Boyce M, Steele IA, Campbell F, Varro A, Pritchard DM. Netazepide, a gastrin receptor antagonist, normalises tumour biomarkers and causes regression of type 1 gastric neuroendocrine tumours in a nonrandomised trial of patients with chronic atrophic gastritis. PLoS One. 2013 Oct 1;8(10):e76462. doi: 10.1371/journal.pone.0076462. eCollection 2013. PMID 24098507